CLINICAL TRIAL: NCT05870189
Title: Remotely Delivered Cognitive Multisensory Rehabilitation for Sensory and Motor Recovery After Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMR
Record Dates: First submitted 2023-04-28; First posted 2023-05-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote CMR (Experimental): adults with SCI without restriction for race, sex or socio-economic status randomized to CMR intervention.
  Interventions: Behavioral: Remote CMR
- Remote exercises (Placebo Comparator): adults with SCI without restriction for race, sex or socio-economic status randomized to remote exercise intervention.
  Interventions: Behavioral: Remote Exercise

INTERVENTIONS:
Behavioral: Remote CMR — 12 weeks of remote CMR is done 3x/week, 45 min/session.
  Arms: Remote CMR
Behavioral: Remote Exercise — 12 weeks of remote exercise is done 3x/week, 45 min/session.
  Arms: Remote exercises

SUMMARY:
So far, therapies have limited success in functional recovery in adults with chronic SCI. By introducing remote cognitive multisensory rehabilitation (CMR), which has shown significant functional improvements due to neurological recovery when delivered in-person, transformative results that (i) provide a potentially effective new therapy within the healthcare system, accessible to more patients, and (ii) demonstrate brain function changes alongside improved function in chronic SCI are anticipated. The results will inform and justify a large scale federally funded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old, with an incomplete or complete SCI/D of ≥ 3months, medically stable.
* be recruited from Hospitals within the Minnesota Regional Spinal Cord Injury Model System (MN Regional SCIMS), HealthPartners Neuroscience Center, Minneapolis VA Healthcare System, Duluth, and in the community.

Exclusion Criteria:

* adults with MRI contra-indications (stabilizing hardware is typically MRI safe);
* adults with uncontrolled seizure disorder;
* adults with cognitive impairment and/or communicative disability (e.g., due to brain injury) that prevent them from following directions or from learning;
* adults with with ventilator dependency;
* adults with other major medical complications
* pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Neurologic Exam | baseline
  a clinical test originally designed to describe the extent and severity of a patient's SCI/D
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Neurologic Exam | 12 weeks
  a clinical test originally designed to describe the extent and severity of a patient's SCI/D
the Neuromuscular Recovery Scale (NRS) | baseline
  includes 11 items focused on the capacity of the trunk and lower extremity muscles to perform tasks such as sit, trunk extension, sit to stand, walking, and step retraining. The NRS provides a functional recovery measure that focuses on non-compensatory recovery.
the Neuromuscular Recovery Scale (NRS) | 12 weeks
  includes 11 items focused on the capacity of the trunk and lower extremity muscles to perform tasks such as sit, trunk extension, sit to stand, walking, and step retraining. The NRS provides a functional recovery measure that focuses on non-compensatory recovery.
The SCI-FI/AT | baseline
  (32 items) reliably measures function in the domains of basic mobility, self-care, fine motor function, and ambulation.
The SCI-FI/AT | 12 weeks
  (32 items) reliably measures function in the domains of basic mobility, self-care, fine motor function, and ambulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States